CLINICAL TRIAL: NCT02966808
Title: Retrospective Study About Long-term Effect of Fampridine in Patients With Multiple Sclerosis
Brief Title: Retrospective Observational Study About Long-term Effect of Fampridine in Patients With Multiple Sclerosis
Acronym: RETROFAM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, María Luisa Martinez Gines, Medical Doctor in Neurology, Hospital General Universitario Gregorio Marañon
Other Study IDs: RETROFAM
Record Dates: First submitted 2016-11-02; First posted 2016-11-17 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinical measures: multiple sclerosis patients in treatment with fampridine
  Interventions: Behavioral: cognitive and behavioural questionnaires

INTERVENTIONS:
Behavioral: cognitive and behavioural questionnaires
  Other Names: PASAT, SDMT, MSQoL-54, MSFIS, T25WF, MSWS12

SUMMARY:
Mobility problems in multiple sclerosis (MS) is a frequent symptom. It might appear in almost 93% of patients in the first 15 years of the disease, being a clear problem for their normal living. Nevertheless, therapeutic options for this symptom are few and optimal for only some patients.

DETAILED DESCRIPTION:
The mechanism of action of fampridine has a direct effect on mobility and it´s based on voltage-dependent potassium channels functioning, causing an improvement of conductivity of action-potential in neurons. This is why nowadays is the only approved drug to treat walking and mobility problems in MS. Results obtained after Phase III randomized clinical trials proved improvement in walking ability measured using the Timed 25 Walking Feet test (T25WF).

There are few studies regarding fampridine effects on symptoms different from mobility. The ENABLE Phase VI study found the first data related with the long-term impact of this treatment in physical and psychological function in patients according to their own perception. Results from this study indicated that, after one year of treatment, patients perceived a sustained benefit in their health, both physical and psychologically.

ELIGIBILITY:
Inclusion Criteria:

* patients with multiple sclerosis with fampridine treatment

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with multiple sclerosis elegible for fampridine treatment according to drug lable.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in speed of processing | change from baseline to 15 days, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months and 36 moths after initiating treatment.
  Symbol Digit Modality Test (SDMT)
change in attention | change from baseline to 15 days, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months and 36 moths after initiating treatment.
  Paced Auditory Serial Addition Test (PASAT)
change in walking ability | change from baseline to 15 days, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months and 36 moths after initiating treatment.
  Timed 25 walking feet (T25WF)
change in perception of walking ability | change from baseline to 15 days, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months and 36 moths after initiating treatment.
  Multiple Sclerosis Walking Scale 12 (MSWS12)

SECONDARY OUTCOMES:
change in fatigue | change from baseline to 15 days, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months and 36 moths after initiating treatment.
  Multiple Sclerosis Fatigue Impact Scale (MSFIS)
change in quality of life | change from baseline to 15 days, 3 months, 6 months, 9 months, 12 months, 18 months, 24 months, 30 months and 36 moths after initiating treatment.
  Multiple Sclerosis Quality of Life 54 (MSQoL-54)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luisa Martínez-Ginés, MD, Principal Investigator — Neurologist
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided